CLINICAL TRIAL: NCT02645552
Title: Pre-hospital Administration of Tranexamic Acid for Adults With Moderate and Severe Traumatic Brain Injury: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Pre-hospital Administration of Tranexamic Acid for Moderate and Severe Traumatic Brain Injury
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai Pudong Emergency Center (Unknown)
Responsible Party: Principal Investigator, Guoyi Gao, Professor, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TXA4TBI
Record Dates: First submitted 2015-12-22; First posted 2016-01-01 (Estimated); Last update posted 2016-01-01 (Estimated); Status verified 2015-12

CONDITIONS: Brain Injuries, Traumatic
Keywords: Traumatic brain injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Tranexamic Acid; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tranexamic acid (Experimental): Focused intervention
  Interventions: Drug: Tranexamic Acid
- Sodium chloride (Placebo Comparator): Placebo control
  Interventions: Other: Sodium chloride

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid 1 gram in 100 ml saline, by intravenous drip over 10 minutes, once patient admitted to the trial on the spot of TBI
  Other Names: Transamin
  Arms: Tranexamic acid
Other: Sodium chloride — Sodium Chloride solution (0.9%) 1 ml (gram) in 100 ml saline, by intravenous drip over 10 minutes, once patient admitted to the trial on the spot of TBI
  Other Names: Placebo
  Arms: Sodium chloride

SUMMARY:
This study is a prospective single-centre randomized trial to compare the effect of tranexamic acid versus placebo in the pre-hospital management of patients with moderate and severe traumatic brain injury.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) remains a significant public health concern with poor outcome and one of the unmet needs in medical care. Tranexamic acid (TXA) has been shown to reduce blood loss after elective surgery and improve outcomes after traumatic injury due to bleeding without obvious adverse events. In the CRASH-2 Intracranial Bleeding Study, with the nested randomized trial design, the study showed that treatment with TXA within 8 hours of injury was associated with a reduction in haemorrhage growth [adjusted difference, -3.8 ml, 95% confidence interval (CI), -11.5 ml to 3.9 ml], fewer focal ischaemic lesions [adjusted odds ratio (OR) 0.54, 95% CI 0.20 to 1.46] and fewer death (adjusted OR 0.49, 95% CI 0.22 to 1.06) for patients with TBI (Glasgow coma score ≤ 14). The study also provided direction for future research of TXA in TBI, especially for the patients with moderate and severe TBI in whom an intracranial intracranial bleed (defined as the presence of parenchymal, subdural or epidural haemorrhage) is common.

Furtherly, results of the CRASH-2 trial stressed the importance of early adminstration with TXA for trauma patients, with the evidence showing that treatment of TXA within 1 hour post injury could significantly reduce the risk of death, while the benefit did not exist when TXA was administered more than 3 hours after injury. If the use of TXA could be incorporated into the pre-hospital management of TBI, the outcome of traumatically injured patients would be improved in an early stage. Thus, our study sets out to employ a randomized controlled study design, with a sample of 400 patients, to evaluate the efficacy and safety of early use of TXA in the pre-hospital management for moderate and severe TBI.

ELIGIBILITY:
Inclusion Criteria:

* moderate to severe injuries(post-resuscitation scores Glasgow coma score of 4-12)
* age >= 18 year
* non-penetrating TBI in 2 hours onset

Exclusion Criteria:

* patients with coagulopathy
* pregnancy
* receiving any medication which affects haemostasis
* no consenting form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Glasgow Outcome Scale (GOS) | 6 months post injury
  The GOS is five-category scale used for assessing the neurologic outcome after brain injury as follows: 1, death; 2, vegetative state - unable to interact with the environment; 3, severe disability - unable to live independently but able to follow commands; 4, moderate disability - capable of living independently but unable to return to work or school; and 5, good recovery - able to return to work or school. In our statistical analyses, the outcome will be further dichotomized in unfavorable (GOS 1-3) vs favorable (GOS 4-5); the proportion of unfavorable outcome will be compared between groups.

SECONDARY OUTCOMES:
Vascular occlusive events | 6 months post injury
  Vascular occlusive events includes myocardial infarction, stroke, pulmonary embolism, clinical evidence of deep vein thrombosis.
Death | 6 months post injury
Length of intensive care unit stay | 6 months post injury

CONTACTS AND LOCATIONS:
Overall Officials: Guoyi Gao, MD, PhD, Principal Investigator — Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University
Locations (1):
- Department of Neurosurgery, Ren Ji Hospital, School of Medicine, Shanghai Jiao Tong University, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] CRASH-2 trial collaborators; Shakur H, Roberts I, Bautista R, Caballero J, Coats T, Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejia-Mantilla J, Miranda J, Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive events, and blood transfusion in trauma patients with significant haemorrhage (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. PMID 20554319